CLINICAL TRIAL: NCT03699566
Title: The Relationship Between Trunk Muscle Endurance, Respiratory Functions and Respiratory Muscle Strength in Healthy Individuals
Brief Title: Assessment of Trunk Muscle Endurance, Respiratory Functions and Respiratory Muscle Strength in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: T.C. Dumlupınar Üniversitesi (Other)
Responsible Party: Principal Investigator, Fuat YÜKSEL, Research assistant, Gazi University
Other Study IDs: Fuat1
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Respiratory Muscles and Core Stabilization
Keywords: Trunk muscle endurance; respiratory muscle strength; respiratory functions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Individuals aged 18-65 without chronic disease.
  Interventions: Assessment of Respiratory Muscle Strength, Spirometer, Trunk Muscles Endurance Tests
  Interventions: Other: Assessment of Respiratory Muscle Strength; Other: Spirometer; Other: Trunk Muscles Endurance Tests

INTERVENTIONS:
Other: Assessment of Respiratory Muscle Strength — The maximal voluntary inspiratory (PImax) and expiratory (PEmax) pressure measurements of the subjects were performed using Cosmed Pony FX model (Italy 2001) while the subjects were in the sitting position with a nose clip.
Other: Spirometer — Spirometric measurements were conducted with Cosmed, Pony FX (descopt spirometer- Italy 2001) spirometer using a nose clips while the subjects were in 90 degree relaxed sitting position.
Other: Trunk Muscles Endurance Tests — Trunk muscle endurance of the subjects was measured using four different tests (Side Bridge Test- SBT, Prone Bridge Test- PBT, Flexor Endurance Test- FET, Sorenson Test- ST).

SUMMARY:
The diaphragm forms the upper segment of the core structure. At the same time, the diaphragm muscle acts as the first muscle in the inspiratory function. The aim of this study was to investigate the relationship between respiratory functions and trunk muscle endurance. In this context, respiratory muscle strengths, respiratory functions and body muscle endurance of the cases were measured.

DETAILED DESCRIPTION:
The study was conducted on 60 healthy volunteers ranging in age from 20 to 36 years. 27 woman and 33 men participated in the study. Respiratory muscle strength, trunk muscle endurance, pulmonary function test values and physical activity levels were evaluated for the subjects participating in the study.Respiratory muscle strength and respiratory function tests were performed with a Cosmed Pony Fx portable spirometer. Trunk muscle endurance of the individuals were evaluated by prone bridge, side bridge, flexor endurance and sorensen test.

ELIGIBILITY:
Inclusion Criteria:

* Not having any chronic disease
* Not being pregnant

Exclusion Criteria:

* History of cardiopulmonary disease.
* Morbid obesity
* Major surgical history

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Maximal voluntary inspiratory (PImax) | Baseline assessment no follow- up
  inspiratory pressure measurement in cm H2O
Prone Bridge Test | Baseline assessment no follow- up
  Trunk endurance test aganist the time

SECONDARY OUTCOMES:
Maximal voluntary expiratory (PEmax) | Baseline assessment no follow- up
  Expiratory pressure measurement in cm H2O
Side Bride Test | Baseline assessment no follow- up
  Trunk endurance test aganist the time
Forced Vital Capacity ( FVC) | Baseline assessment no follow- up
  Dinamic volume measure for lungs
Forced Expiratuar Volume 1. Second ( Fev1) | Baseline assessment no follow- up
  Dinamic volume measure for lungs
Abdominal Flexor Endurance Test | Baseline assessment no follow- up
  Trunk endurance test aganist the time
Sorensen Test | Baseline assessment no follow- up
  Back Muscles endurance test aganist the time

CONTACTS AND LOCATIONS:
Overall Officials: Nevin Güzel, prof. dr., Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided